CLINICAL TRIAL: NCT03317548
Title: Chung Shan Medical University Hospital
Brief Title: A Comparison of Clinical Outcomes of Warmed Embryo Vitrified at 2PN Stage and Fresh Embryo Transfers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yeh, Director of The Institutional Review Board, Chung Shan Medical University
Other Study IDs: CS17064
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Infertility, Female; Reproductive Disorder
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fresh embryo transfer: patients with fresh day 3 embryo transfer after oocyte pick up, the hormone including FSH, LH, E2 and progesterone was test before embryo transfer for analysis. The clinical outcomes including implantation and pregnancy were checked and recorded.
  Interventions: Diagnostic Test: progesterone; Diagnostic Test: day 3 embryo
- frozen embryo transfer: freeze-all embryo was performed after oocyte fertilization, the hormone including FSH, LH, E2 and progesterone was test before oocyte pick up and embryo transfer for analysis.
  vitrification of pronuclear stage embryo (zygote) and frozen embryo transfer
  Interventions: Diagnostic Test: progesterone; Diagnostic Test: day 3 embryo

INTERVENTIONS:
Diagnostic Test: progesterone — according progesterone level to decide fresh or frozen embryo transfer
Diagnostic Test: day 3 embryo — according day 3 embryo to decide fresh or frozen embryo transfer

SUMMARY:
The aim of this study was to compare the clinical outcomes between fresh embryo and frozen embryo transfer in in vitro fertilization (IVF). All frozen embryo was vitrified at pronuclear stage (2PN) and cultured to cleavage embryos for transfer.

This is a retrospective study. All IVF cycles were included in this study and further divided into fresh and frozen embryo transfer groups. The collection data including: stimulation protocols, medicines, blood test results, pregnancy test and all clinical data. The primary outcome is pregnancy rate and secondary outcome is implantation rate.

DETAILED DESCRIPTION:
Study design

Study progress:

Stage 1: collection of all data from frozen embryo transfer and fresh embryo transfer groups.

Stage 2: selection data and check the delivery outcomes Stage 3: analysis data and presentation. Including criteria: all patients who underwent IVF. Excluding criteria: No. Statistics analysis: chi-test, t-test

Assessment point:

Primary endpoint: pregnancy rate Secondary endpoint: implantation rate Withdraw criteria: not application. Treatments: not application. Collection number: 500 patients. Scheduled trial period: 2017.05.01~2018.04.30

Expected research results:

The implantation rate in frozen embryo transfer group which vitrified at 2PN stage is higher than fresh embryo transfer.

The pregnancy rate in frozen embryo transfer group which vitrified at 2PN stage is higher than fresh embryo transfer.

This study is only data analysis, no additional collection of samples. This study does not involve vulnerable groups.

ELIGIBILITY:
Inclusion Criteria:

* all patients with in vitro fertilization protocols

Exclusion Criteria:

* none

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all patients underwent in vitro fertilization protocols in Lee Women's Hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | HCG test at day 15 after embryo transfer or day 18 after oocyte pick up
  HCG test

CONTACTS AND LOCATIONS:
Overall Officials: Maw-Shang Lee, Phd, Study Chair — Lee Women's Hospital
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided